CLINICAL TRIAL: NCT03479671
Title: A Dose Finding Study for Fat-Induced Insulin Resistance in Healthy Volunteers
Brief Title: Low Dose Fat-Induced Insulin Resistance
Acronym: BCAA
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Zoltan Arany, Associate Professor Of Medicine, University of Pennsylvania
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 831425
Record Dates: First submitted 2018-03-20; First posted 2018-03-27 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Diabetes Mellitus, Type 2; Insulin Resistance; Insulin Sensitivity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — soybean oil, phospholipid emulsion

STUDY DESIGN:
Intervention Model Description: Baseline insulin sensitivity will be measured in healthy volunteers, and then 1-3 weeks later insulin sensitivity will be measured in response to a low-dose fatty acid infusion. If there is no response to this low-dose infusion, then 1-3 weeks later insulin sensitivity will be measured in response to a medium-dose fatty acid infusion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Saline (No Intervention): Insulin sensitivity (rate of glucose disposal)
- Low Dose Fatty Acids (Experimental): Insulin sensitivity (rate of glucose disposal) in response to 30 ml/hr fatty acid infusion
  Interventions: Drug: Intralipid, 20% Intravenous Emulsion
- Medium Dose Fatty Acids (Experimental): Insulin sensitivity (rate of glucose disposal) in response to 60 ml/hr fatty acid infusion
  Interventions: Drug: Intralipid, 20% Intravenous Emulsion

INTERVENTIONS:
Drug: Intralipid, 20% Intravenous Emulsion — Fatty Acid Infusion, either in low-dose (30 ml/hr) or medium-dose (60 ml/hr)
  Arms: Low Dose Fatty Acids; Medium Dose Fatty Acids

SUMMARY:
The primary goal of this study is to determine the dose of fatty acids that acutely induces mild insulin resistance in healthy volunteers. We hypothesize that a low-dose of fatty acid infusion (Intralipid/heparin) will cause a mild insulin resistance. The dose of fatty acid infusion that reliably causes mild insulin resistance will be selected for use in future studies.

DETAILED DESCRIPTION:
This study is designed to test the hypothesis that a low-dose of fatty acid infusion (Intralipid/heparin) will cause mild insulin resistance. This dose-finding study is critical for future studies on free-fatty acid induced insulin resistance.

Healthy male and healthy female volunteers will undergo a 6 hour hyperinsulinemic-euglycemic clamp, in order to establish insulin sensitivity parameters in the presence of fatty acid co-infusion. The subjects will then return 1-3 weeks later, and undergo another 6 hour HIE clamp, this time in the presence of low-dose fatty acid co-infusion (30ml/hr). If this dose does not achieve ~25% reduction in the rate of glucose disposal, then the dose-confirmation study will be repeated 1-3 weeks later with a medium-dose fatty acid co-infusion (60ml/hr).

A dose-response effect of fatty acids on insulin resistance has been demonstrated before, but not in the precise conditions of our study. This dose-finding study is critical because future studies require a reliable dose of fatty acid infusion, and the exact dose of fatty acid infusion that causes mild insulin resistance may be different in the conditions of our study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are able to provide written informed consent and to comply with the procedures of the study protocol

Exclusion Criteria:

* History of diabetes
* History of diabetes in more than one first-degree relative
* Body mass index (BMI) <19 or >27 kg/m2
* HbA1c >5.7%
* Blood Pressure: systolic >160 mmHg or diastolic > 100 mmHg
* Baseline hemoglobin concentration < 11 g/dl in women and < 12 g/dl in men
* Estimated glomerular filtration rate < 55 ml/min/1.73 m2 (calculated using the subject's measured serum creatinine and the Modification of Diet in Renal Disease [MDRD] study estimation formula).
* Presence of soy or egg allergies (due to possible reactions with fat infusate)
* For female participants: Positive pregnancy test, presently breast-feeding, or unwillingness to use effective contraceptive measures for the duration of the study. Oral contraceptives, Norplant®, Depo-Provera®, and barrier devices with spermicide are acceptable contraceptive methods; condoms used alone are not acceptable.
* Known active alcohol or substance abuse
* Use of tobacco within the previous year
* Severe co-existing cardiac disease, characterized by any one of these conditions:

  1. history of myocardial infarction within past 6 months;
  2. history of ischemia on functional cardiac exam within the last year;
  3. history of left ventricular ejection fraction < 30%.
* Persistent elevation of liver function tests > 1.5 times normal upper limits
* Hyperlipidemia (fasting LDL cholesterol > 130 mg/dl, treated or untreated; and/or fasting triglycerides > 200 mg/dl)
* Receiving treatment for a medical condition requiring chronic use of systemic steroids, except for the use of ≤ 5 mg prednisone daily, or an equivalent physiological dose of hydrocortisone
* Presence of a seizure disorder
* Use of any investigational agents within 4 weeks of enrollment
* Any medical condition, which in the opinion of the investigator, will interfere with the safe completion of the study
* History of pancreatitis
* Presence of a metal allergy (aluminum)

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male or Female at birth.
Enrollment: 12 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Insulin Sensitivity | 6 hours
  Rate of Glucose Disposal (mg/kg/min)

CONTACTS AND LOCATIONS:
Overall Officials: Zoltan P Arany, MD, PhD, Principal Investigator — Associate Professor of Medicine
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided